CLINICAL TRIAL: NCT02516514
Title: The Only Blood Culture for Diagnosis of Bacteremia - Comparative Study of Practice
Acronym: HEMU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-033
Record Dates: First submitted 2015-07-28; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Bloodstream Infection
Keywords: Blood culture; Bacteremia; Single sampling
MeSH Terms: conditions — Sepsis; Bacteremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-sampling strategy (Experimental): 2 or 3 blood cultures in 24 hours worked at ½ hour intervals with seeding at least a pair of flasks, aerobic and anaerobic, by blood culture.
  Interventions: Procedure: Single-sampling strategy vs multi-sampling strategy for the diagnosis of bacteremia
- Single-sampling strategy (Active Comparator): 1 single dose of venous blood 30ml ± 10ml with seeding 4 blood culture bottles (aerobic and anaerobic 2 2).
  Interventions: Procedure: Single-sampling strategy vs multi-sampling strategy for the diagnosis of bacteremia

INTERVENTIONS:
Procedure: Single-sampling strategy vs multi-sampling strategy for the diagnosis of bacteremia — Comparison between two strategies of blood culture (single-sampling strategy and multi-sampling strategy) for the diagnosis of bacteremia

SUMMARY:
Current recommendations for the diagnosis of bacteremia based on the embodiment February-March blood cultures separated by a minimum interval of 30 minutes. Each blood culture comprises seeding a pair of aerobic and anaerobic vials inoculated each with 5 to 10 ml of blood. The sensitivity and specificity of this technique depends essentially on the amount of blood removed since there is a direct relationship between the volume of blood inoculated into each flask and the efficiency of the technique. A preliminary study conducted at the University Hospital of Caen found that 14-30% of patients depending on the services had received only one blood culture. In addition, at least four blood cultures in 24 hours were taken for 10 to 20% of patients. The practice of a single blood culture reduces the sensitivity of the analysis due to insufficient total amount of blood collected. The practice of too many blood cultures increases the risk of false positive (presence of contaminating bacteria), generates extra work for healthcare personnel (and laboratory) and represents a significant cost for an unproven benefit.

The investigators propose to evaluate a single blood culture sampling technique with seeding 4 vials (2 aerobic and anaerobic 2).

DETAILED DESCRIPTION:
Blood cultures will be collected from patients admitted with on of the following signs: fever (≥38.5°C), hypothermia (≤36°C), chills or shock. For the first blood culture, 40 mL of blood will be obtained aseptically by a single phlebotomy and equally distributed into two BacT/Alert FA aerobic bottles and two BacT/Alert FN anaerobic bottles (bioMérieux, La-Balme-les-Grottes, France). The four bottles will be labelled from one to four in the following order: aerobic-anaerobic-aerobic-anaerobic. Within the next 24 h, one to three other 20-mL blood cultures consisting of a single pair of aerobic and anaerobic bottles will have to be performed, spaced by a minimum of 30 minutes. Bottles will be incubated for 5 days or until positivity reported by the BacT/Alert 3D instrument.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is at least 18 years
* Patients admitted to an emergency department of a three CHU Caen, Lille, Rouen
* Patient with clinical justifying the realization of blood cultures (as good practice recommendations)
* Patients who received information about the study or if his legal representatives or his close entourage
* Patient not objecting to the venipuncture

Exclusion Criteria:

* Patient who direct venipuncture is impossible
* Patient refusing venipuncture
* Patient aged under 18
* Patient with impaired vigilance and not accompanied by a family member or a trusted person may receive clear information protocol
* Vulnerable Patient and not accompanied by a family member or a trusted person may receive clear information protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Rate of pathogens identified by each strategy | baseline

SECONDARY OUTCOMES:
Proportion of blood cultures contaminated in each strategy | baseline

REFERENCES:
- [Background] Cockerill FR 3rd, Wilson JW, Vetter EA, Goodman KM, Torgerson CA, Harmsen WS, Schleck CD, Ilstrup DM, Washington JA 2nd, Wilson WR. Optimal testing parameters for blood cultures. Clin Infect Dis. 2004 Jun 15;38(12):1724-30. doi: 10.1086/421087. Epub 2004 May 25. PMID 15227618
- [Background] Li J, Plorde JJ, Carlson LG. Effects of volume and periodicity on blood cultures. J Clin Microbiol. 1994 Nov;32(11):2829-31. doi: 10.1128/jcm.32.11.2829-2831.1994. PMID 7852579
- [Background] Arendrup M, Jensen IP, Justesen T. Diagnosing bacteremia at a Danish hospital using one early large blood volume for culture. Scand J Infect Dis. 1996;28(6):609-14. doi: 10.3109/00365549609037969. PMID 9060065
- [Background] Lamy B, Roy P, Carret G, Flandrois JP, Delignette-Muller ML. What is the relevance of obtaining multiple blood samples for culture? A comprehensive model to optimize the strategy for diagnosing bacteremia. Clin Infect Dis. 2002 Oct 1;35(7):842-50. doi: 10.1086/342383. Epub 2002 Sep 10. PMID 12228821
- [Background] Lee A, Mirrett S, Reller LB, Weinstein MP. Detection of bloodstream infections in adults: how many blood cultures are needed? J Clin Microbiol. 2007 Nov;45(11):3546-8. doi: 10.1128/JCM.01555-07. Epub 2007 Sep 19. PMID 17881544